CLINICAL TRIAL: NCT00001878
Title: Contribution of Insulin-Like Growth Factor-I (IGF-I) and Its Binding Protein (IGFBP3) to Increased Left Ventricular Mass in Familial Hypertrophic Cardiomyopathy Caused by Distinct Sarcomeric Mutations
Brief Title: Factors Contributing to Increased Left Ventricle Size in Patients With Abnormally Enlarged Hearts
Status: Completed | Type: Observational
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 990058; 99-H-0058
Record Dates: First submitted 1999-11-03; First posted 1999-11-04 (Estimated); Last update posted 2008-03-04 (Estimated); Status verified 2002-08

CONDITIONS: Hypertrophic Cardiomyopathy; Left Ventricular Hypertrophy
Keywords: Growth Hormone; Cardiac Hypertrophy; Hypertrophic Cardiomyopathy; Sarcomeric Gene Mutations
MeSH Terms: conditions — Cardiomyopathy, Hypertrophic; Hypertrophy, Left Ventricular; Cardiomegaly

SUMMARY:
The human heart is divided into four chambers. One of the four chambers, the left ventricle, is the chamber mainly responsible for pumping blood out of the heart into the circulation. There is an inherited condition affecting the heart, passed on through genetics, hypertrophic cardiomyopathy (HCM). HCM causes the left ventricle to become abnormally enlarged (left ventricular hypertrophy LVH).

Some patients with the abnormal genes that may cause HCM do not have the characteristic LVH. Approximately 20 - 40% of patients with the genetic abnormality (missense mutation of genes encoding for sarcomeric protein) actually have an enlarged left ventricle. Because of this, researchers believe there may be other factors, along with the genetic abnormality that contribute to the development of HCM. Researchers are interested in learning more about several factors they suspect may play a role in the development of HCM.

Specifically, researchers plan to study levels of a hormone and the protein it attaches to, which may contribute to the development of an abnormally enlarged heart. Insulin-like growth factor (IGF-1) and insulin-like growth factor binding protein (IGFBP) work together with growth hormone (GH) in the development and maturation of many organ systems. Previous studies have suggested that these hormones affect the development and function of the heart.

Patients participating in this study will undergo a variety of tests including collection of blood samples, echocardiogram of the heart, treadmill exercise test, and continuous electrical monitoring of heart activity (Holter monitor).

DETAILED DESCRIPTION:
Hypertrophic cardiomyopathy (HCM) is a genetic disease with an autosomal dominant pattern of inheritance which is characterized by left ventricular hypertrophy (LVH). HCM is often caused by missense mutations of genes that encode for sarcomeric proteins. The LVH varies markedly in patients with identical sarcomeric gene mutations, and notably, 20 to 40% of subjects with disease mutation do not have LVH as assessed by echocardiography. These findings suggest that other factors affect LV wall thickness in HCM. We wish (1) to investigate the potential role of IGF-I and its binding protein, IGFBP3, in determining increased LV mass in HCM caused by sarcomeric mutations; and (2) to assess myocardial ultrasound backscatter, exercise tolerance, and propensity to arrhythmias, in subjects who have inherited sarcomeric mutations but who do not have LVH.

ELIGIBILITY:
INCLUSION CRITERIA

HCM subjects 5 years or older, with distinct sarcomeric gene mutations and LV wall thickness greater than 15 mm in subjects older than 18 years, and greater than 2 SDs in subjects 18 years of age or younger, as assessed by MRI.

Age- and gender-matched blood relatives with sarcomeric gene mutations but without LVH.

Age- and gender-matched blood relatives without sarcomeric gene mutations.

EXCLUSION CRITERIA

History of hypertension (basal systolic and diastolic pressures above 170 mm Hg and 95 mm Hg, respectively) or another systemic or cardiac disease that may cause cardiac hypertrophy.

History of recent acute illness or other chronic illness that might affect plasma levels of IGF-I and IGFBP3.

History of thyrotoxicosis, diabetes mellitus or abnormally elevated fasting blood sugar.

Any conditions which would exclude patients from undergoing MRI scan.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 175
Dates: Start 1999-02; Study Completion 2002-08

CONTACTS AND LOCATIONS:
Locations (1):
- National Heart, Lung and Blood Institute (NHLBI), Bethesda, Maryland, United States

REFERENCES:
- [Background] Jarcho JA, McKenna W, Pare JA, Solomon SD, Holcombe RF, Dickie S, Levi T, Donis-Keller H, Seidman JG, Seidman CE. Mapping a gene for familial hypertrophic cardiomyopathy to chromosome 14q1. N Engl J Med. 1989 Nov 16;321(20):1372-8. doi: 10.1056/NEJM198911163212005. PMID 2811944
- [Background] Rayment I, Holden HM, Sellers JR, Fananapazir L, Epstein ND. Structural interpretation of the mutations in the beta-cardiac myosin that have been implicated in familial hypertrophic cardiomyopathy. Proc Natl Acad Sci U S A. 1995 Apr 25;92(9):3864-8. doi: 10.1073/pnas.92.9.3864. PMID 7731997
- [Background] Thierfelder L, Watkins H, MacRae C, Lamas R, McKenna W, Vosberg HP, Seidman JG, Seidman CE. Alpha-tropomyosin and cardiac troponin T mutations cause familial hypertrophic cardiomyopathy: a disease of the sarcomere. Cell. 1994 Jun 3;77(5):701-12. doi: 10.1016/0092-8674(94)90054-x. PMID 8205619